CLINICAL TRIAL: NCT01332682
Title: Resistance Training and Physical Functioning in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCCI-09-001-A; SCRIHS 07-164 (Other Grant/Funding Number: EAM 2009)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Cancer; Pharyngeal Cancer; Laryngeal Cancer
Keywords: head and neck cancer; resistance training; nutrition counseling; pharyngeal or laryngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Nutritional Status; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance Training and Nutrition Counseling (Experimental)
  Interventions: Behavioral: Resistance Training and Nutrition Counseling
- Nutrition Counseling (Other)
  Interventions: Behavioral: Nutrition Counseling

INTERVENTIONS:
Behavioral: Nutrition Counseling — Patients will meet once per week with dietitian for the first 6 weeks in 60 minute sessions. Dietitian will telephone each patient weekly for the final 6 weeks of counseling and support.
  Other Names: nutrition
  Arms: Nutrition Counseling
Behavioral: Resistance Training and Nutrition Counseling — Patient will meet with an exercise specialist once per week for the first 6 weeks. Patient will receive guidance in a safe and appropriate exercise regimen based on specific medical history and preference. An exercise specialist will telephone weekly for consultation and support once per week for the final 6 weeks. Also, patient will meet once per week with dietitian for the first 6 weeks in 60 minute sessions. Dietitian will telephone each patient weekly for the final 6 weeks of counseling and support.
  Arms: Resistance Training and Nutrition Counseling

SUMMARY:
The purpose of this feasibility study is to examine the safety and effect of resistance training on muscle strength, lean body mass, physical functioning, fatigue, and quality of life in head and neck cancer patients receiving radiation therapy.

DETAILED DESCRIPTION:
Head and neck cancer (HNCa) patients often lose significant body weight and lean mass which is associated with higher mortality, greater fatigue, poorer quality of life, and reduced physical functioning. Because nutritional supplementation may not consistently improve lean body mass, resistance training may be beneficial. HNCa patients experience unique side effects that impact nutritional status, limiting generalization of exercise intervention study results in other cancer types to HNCa patients. Therefore, 44 HNCa patients will be enrolled in a randomized controlled trial with the following study aims:

Primary study aim: Because this pilot proposal is among the first to attempt a randomized controlled exercise trial in HNCa patients, the primary study aim examines safety and feasibility (e.g., study acceptance, recruitment, intervention process evaluation, adherence, adverse events, retention). The investigators hypothesize that study procedures will require minor alterations in future studies.

Secondary study aim #1: Because effect sizes are necessary for planning efficacy trials, the proposal will compare the effect of a 12-week resistance training plus nutritional counseling intervention versus nutritional counseling alone on muscle strength, lean body mass, physical functioning, fatigue, and quality of life in HNCa patients receiving radiation with or without chemotherapy. The investigators hypothesize that patients receiving resistance training with nutritional counseling will demonstrate greater improvements in the outcomes when compared with participants receiving nutritional counseling alone.

Secondary study aim #2: To enhance adherence in future intervention trials, this proposal will determine resistance training and nutritional adherence rates and associated factors among HNCa patients using attendance records, exercise logs, diet records, self-administered survey, and medical record review. The investigators hypothesize that adherence rates will be lower than that of other cancer populations with correlates including demographic, medical, and psychosocial factors.

Assessments will occur at baseline (first week of radiation), week 6 (mid-intervention), and week 12 (post-intervention). Qualitative and quantitative (e.g., rates, 95% confidence intervals) will assess feasibility and mixed model ANOVA will examine group differences. This information is critical for the design of future resistance training efficacy trials in HNCa patients to prevent lean body mass loss in HNCa patients, potentially reducing mortality, minimizing fatigue, and improving physical functioning and quality of life.

ELIGIBILITY:
Inclusion criteria:

* cancer of the oral cavity, pharynx, larynx, nasal cavity/sinuses, or salivary gland
* ≥ 18 years of age
* English speaking
* radiation therapy planned or underway < 1 week, and
* able to stand

Exclusion Criteria:

* dementia or organic brain syndrome
* severe emotional distress
* active schizophrenia
* quadriplegia or loss of use of limbs or torso
* tendon rupture
* muscle tear
* cancer recurrence
* another diagnoses of cancer in the past 5 years, and
* oncologist refuses to allow screening for possible study participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
safety of head and neck cancer patients | daily (up to 12 weeks)
  adverse events

SECONDARY OUTCOMES:
change in muscle strength | baseline, week 6, and week 12
  dynamometer measurement
Number of patients who adhere to cohort activity schedule | baseline, week 6, and week 12
  completion of exercise or diet recommendations
change in lean body mass | baseline, week 6, week 12
  bioelectrical impedence
change in physical functioning | baseline, week 6, week 12
  physical performance by doing a semi-tandem, tandem, or side by side stance with the feet, an 8 foot walk time, and 5 chair rise and sits
change in fatigue level | baseline, week 6, week 12
  13-item Functional Assessment of Cancer Therapy-Fatigue scale
change in quality of life | baseline, week 6, week 12
  37-item Functional Assessment of Cancer Therapy-Head and Neck scale
Number of head and neck cancer patients recruited to participate | up to 16 months
  to test the feasibility of a randomized controlled exercise trial in head and neck cancer patients receiving radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q Rogers, MD, MPH, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Rogers LQ, Rao K, Malone J, Kandula P, Ronen O, Markwell SJ, Courneya KS, Robbins KT. Factors associated with quality of life in outpatients with head and neck cancer 6 months after diagnosis. Head Neck. 2009 Sep;31(9):1207-14. doi: 10.1002/hed.21084. PMID 19360748
- [Background] Rogers LQ, Malone J, Rao K, Courneya KS, Fogleman A, Tippey A, Markwell SJ, Robbins KT. Exercise preferences among patients with head and neck cancer: prevalence and associations with quality of life, symptom severity, depression, and rural residence. Head Neck. 2009 Aug;31(8):994-1005. doi: 10.1002/hed.21053. PMID 19340875
- [Result] Rogers LQ, Anton PM, Fogleman A, Hopkins-Price P, Verhulst S, Rao K, Malone J, Robbs R, Courneya KS, Nanavati P, Mansfield S, Robbins KT. Pilot, randomized trial of resistance exercise during radiation therapy for head and neck cancer. Head Neck. 2013 Aug;35(8):1178-88. doi: 10.1002/hed.23118. Epub 2012 Jul 30. PMID 22847995